CLINICAL TRIAL: NCT05055388
Title: Epidemiological Investigation of Sepsis in Obstetrics Admitted to ICU From 2008 to 2016 in Beijing China: A First Multicenter Report
Brief Title: Epidemiological Investigation of Sepsis in Obstetrics Admitted to ICU
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Zhiling, Deputy chief doctors, Peking University Third Hospital
Other Study IDs: LM2020443
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Maternal Sepsis; Intensive Care Units; Drug Resistance, Multiple
MeSH Terms: conditions — Pregnancy Complications, Infectious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group with sepsis complicated with multidrug-resistant bacteria: Obstetrics diagnosed with sepsis were divided to group with sepsis complicated with multidrug-resistant bacteria if microbial culture results showed multidrug-resistance.
  Interventions: Other: Multidrug-resistant bacteria
- Group with sepsis complicated with none multidrug-resistant bacteria: Obstetrics diagnosed with sepsis were divided to group with sepsis complicated with none multidrug-resistant bacteria if microbial culture results showed none-multidrug-resistance or no positive result of microbial culture.

INTERVENTIONS:
Other: Multidrug-resistant bacteria — Multidrug resistance was defined as acquired non-susceptibility to at leas one agent in three or more antimicrobial categories.
  Groups: Group with sepsis complicated with multidrug-resistant bacteria

SUMMARY:
Sepsis is still the main cause of maternal death, accounting for 11% of maternal deaths. Early identification of high risk factors of sepsis and early intervention can improve the prognosis of pregnant women with sepsis. At present, there is no epidemiological investigation report on sepsis in ICU in China.

DETAILED DESCRIPTION:
Although great progress has been made in maternal care in China in recent years, the maternal mortality rate in China has remained high in the past three years, fluctuating from 19.6-20.1/100000, and there is still a large gap between China and developed countries (12.1/100000). Sepsis is still the main cause of maternal death, accounting for 11% of maternal deaths; Early identification of high risk factors of sepsis and early intervention can improve the prognosis of pregnant women with sepsis. At present, there is no epidemiological investigation report on sepsis in ICU in China. A total of 160 cases of maternal sepsis with ICU admission in any trimester of pregnancy or within 42 days of delivery were reviewed between January 1, 2008, and December 31, 2019. The demographic data including age and gestational age, mode of delivery, the maximal SOFA score, invasive operation before sepsis, sepsis focuses, intervention, microbial culture results, body temperature and blood routine were reviewed to investigate the incidence and mortality of maternal sepsis in intensive care unit, as well as the incidence of multidrug-resistant bacteria and the risk factors of multidrug resistance.

ELIGIBILITY:
Inclusion Criteria: Obstetrics with sepsis in any trimester of pregnancy or within 42 days of delivery -

Exclusion Criteria: The electronic medical record is lost. Patients with incomplete infection data: if the temperature sheet is ambiguous and the temperature data is not recorded in the medical record.

-

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obstetrics with sepsis in any trimester of pregnancy or within 42 days of delivery
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of Maternal sepsis in intensive care unit | January 2008 to December 2019
  The incidence of Maternal sepsis in ICU represents as proportion based on the total number of of maternal ICU admissions and is expressed per 100 deliveries.
Sepsis related maternal mortality | January 2008 to December 2019
  Sepsis related maternal mortality in hospitals represents as proportion based on the total number of maternal sepsis in intensive care units and is expressed per 100,000 deliveries.
The incidence of multidrug resistance | January 2008 to December 2019
  The incidence of multidrug resistance represents as proportion based on the total number of of maternal sepsis in ICU and is expressed per 100 deliveries. Multidrug resistance was defined as acquired non-susceptibility to at leas one agent in three or more antimicrobial categories.

SECONDARY OUTCOMES:
The length of ICU stay | January 2008 to December 2019
  The date of transferring to wards or death minus the date of ICU admission
Hospital length | January 2008 to December 2019
  Discharge date minus admission date

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No